CLINICAL TRIAL: NCT02601053
Title: The Fear F8ctor Study - Does Fear Induce a Blood Curdling State? The Origin Behind the Phrase Unravelled
Brief Title: The Fear F8ctor Study - Does Fear Induce a Blood Curdling State?
Acronym: FF8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, B.Nemeth, MD, Leiden University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P15.146; NL53805.058.15 (Other: Central Committee on Research Involving Human Subjects)
Record Dates: First submitted 2015-11-05; First posted 2015-11-10 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Blood Coagulation Disorder
MeSH Terms: conditions — Blood Coagulation Disorders | interventions — Motion Pictures; Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dull (boring) movie (Active Comparator): Participants will be exposed to a dull (i.e. boring) movie followed by a scary (i.e. horrifying) movie.
  Interventions: Other: Dull movie; Other: Scary (horrifying) movie; Other: Heart rate measurement
- Scary (horrifying) movie (Experimental): Participants will be exposed to a scary (i.e. horrifying) movie followed by a to a dull (i.e. boring) movie.
  Interventions: Other: Dull movie; Other: Scary (horrifying) movie; Other: Heart rate measurement

INTERVENTIONS:
Other: Dull movie — A dull movie (duration approximately 90 minutes)
Other: Scary (horrifying) movie — A scary movie (duration approximately 90 minutes)
Other: Heart rate measurement — Heart rate measurement using a actiheart device

SUMMARY:
For centuries the term "blood curling" has been used to describe extreme frightening situations. However, the origin of this ancient theory has never been studied and it remains unknown if fear induces the coagulation system.The objective was to explore the effects of acute fear on the coagulation system while sitting still. In a crossover study design healthy subjects will be exposed to a horrifying e.g. scary movie followed by a dull e.g. flat movie which is shown at least 1 week after the first movie on the same day of the week at the same time of the day. Participants will be recruited among students from the Leiden University Medical Center. Blood will be drawn from the cubital vein 10 minutes before the first movie, directly after the first movie. The same will be done 10 minutes before and directly after the second movie. Blood is drawn by using a needle puncture.

Individual markers of coagulation activity will be determined from the blood samples. Pulse rates will be measured and an anxiety/fear score will be collected from each student for both movies.

DETAILED DESCRIPTION:
Rationale: For centuries the term "blood curling" has been used to describe extreme frightening situations. The term dates back to the medieval physiology, it was believed that the human body contained four chief fluids, blood, phlegm, bile and black bile. It was thought that fear or horror would 'run the blood cold' or 'curdle' (solidify). To date large parts of the complex mechanism of the coagulation cascade have been unravelled and many risk factors for clotting, i.e., thrombosis have been identified. However, the origin of this ancient theory has never been studied and it remains unknown if fear induces the coagulation system.

Objective: To explore the effects of acute fear on the coagulation system while sitting still.

The investigators will compare systemic coagulation markers before and after both movies in each subject: 13 subjects will be exposed to the horrifying movie first, followed by the dull movie (at least 1 week later). Both movies will be shown on the same day of the week, at the same time of the day and will last approximately 90 minutes. One group of 13 will first view the horrifying movie, followed by the dull move the next week (Group I) and 13 subjects will be exposed to the dull movie first, followed by the horrifying movie (Group II). Spacious seats will be used to avoid the effect of immobilisation due to tight cinema seats. Blood is drawn at four time points (TP); (0) before the first movie (baseline), after the first movie (1), before the second movie (2) and after the second movie (3). A needle puncture is used to collect 12 ml of blood at each time point.

Individual markers of coagulation activity will be determined from the blood samples. Pulse rates will be measured and an anxiety/fear score will be collected from each student for both movies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 30 years old
* No medication and otherwise healthy

Exclusion Criteria:

* Any coagulation disorder
* Hormonal anticonception (excluding intrauterine devices)
* Pregnancy or puerperium
* History of Venous thrombosis
* Major surgery or cast immobilisation in the past two months
* Neoplasm or inflammatory disease

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in Factor VIII:C (mean change before and after movie) between movies | Four time points (TP); (0) before the first movie (baseline), after the first movie [90 minutes](1), before the second movie (baseline, 2) and after the second movie [90 minutes](3). All blood will be drawn within 15 minutes before or after the movie.
  The mean change in FVIII:C (in IU/dL) levels after seeing a scary movie (ie from timepoint 0 to 1 in study arm I and from timepoint 2 to timepoint 3 for treatment arm II will be compared to the mean change after seeing a dull movie. A paired student t-test is used to compare the two mean changes in coagulation markers.
Change in D-dimer (mean change before and after movie) between movies | Four time points (TP); (0) before the first movie (baseline), after the first movie [90 minutes](1), before the second movie (baseline, 2) and after the second movie [90 minutes](3). All blood will be drawn within 15 minutes before or after the movie.
  The mean change in D-dimer(in ng/mL) levels after seeing a scary movie (ie from timepoint 0 to 1 in study arm I and from timepoint 2 to timepoint 3 for treatment arm II will be compared to the mean change after seeing a dull movie. A paired student t-test is used to compare the two mean changes in coagulation markers.
Change in Thrombin and Antithrombin complexes (TATc) (mean change before and after movie) between movies | Four time points (TP); (0) before the first movie (baseline), after the first movie [90 minutes](1), before the second movie (baseline, 2) and after the second movie [90 minutes](3). All blood will be drawn within 15 minutes before or after the movie.
  The mean change in TATc (in mcg/L) levels after seeing a scary movie (ie from timepoint 0 to 1 in study arm I and from timepoint 2 to timepoint 3 for treatment arm II will be compared to the mean change after seeing a dull movie. A paired student t-test is used to compare the two mean changes in coagulation markers.
Change in Prothrombin fragments 1+2 (F1+2) (mean change before and after movie) between movies | Four time points (TP); (0) before the first movie (baseline), after the first movie [90 minutes](1), before the second movie (baseline, 2) and after the second movie [90 minutes](3). All blood will be drawn within 15 minutes before or after the movie.
  The mean change in F1+2 (in umol/dL) levels after seeing a scary movie (ie from timepoint 0 to 1 in study arm I and from timepoint 2 to timepoint 3 for treatment arm II will be compared to the mean change after seeing a dull movie. A paired student t-test is used to compare the two mean changes in coagulation markers.

SECONDARY OUTCOMES:
Difference of Heart Rate (peaks in heart rate) between movies | During the entire movie the heart rate is recorded [up to 90 minutes]. Heart rate peaks (above average) will be compared between movies in one individual.
  Heart rates will be measures in beats per minute during the entire movie, using an actiheart device that monitores the heart rate every 15 seconds.
Difference of the Visual Analogue Scale on Fear between movies | VAS scale, directly after dull movie [90 minutes] and directly after scary movie [90 minutes] for each individual
  A VAS (0-10 points) on fear is recorded from every participant after they have seen the dull and scary movie.

CONTACTS AND LOCATIONS:
Overall Officials: Banne Nemeth, MD, Principal Investigator — Leiden University Medical Center

REFERENCES:
- [Derived] Nemeth B, Scheres LJ, Lijfering WM, Rosendaal FR. Bloodcurdling movies and measures of coagulation: Fear Factor crossover trial. BMJ. 2015 Dec 16;351:h6367. doi: 10.1136/bmj.h6367. PMID 26673787